CLINICAL TRIAL: NCT01325350
Title: Safety and Efficacy Study of Bimatoprost in the Treatment of Women With Female Pattern Hair Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192024-058; 2011-000380-27 (EudraCT Number)
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-03

CONDITIONS: Alopecia; Baldness
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- bimatoprost Formulation A (Experimental): Approximately one mL dose applied evenly onto pre-specified area on scalp, once daily for 6 months.
  Interventions: Drug: bimatoprost Formulation A
- bimatoprost Formulation B (Experimental): Approximately one mL dose applied evenly onto pre-specified area on scalp, once daily for 6 months.
  Interventions: Drug: bimatoprost Formulation B
- bimatoprost Formulation C (Experimental): Approximately one mL dose applied evenly onto pre-specified area on scalp, once daily for 6 months.
  Interventions: Drug: bimatoprost Formulation C
- bimatoprost vehicle solution (Placebo Comparator): Approximately one mL dose applied evenly onto pre-specified area on scalp, once daily for 6 months.
  Interventions: Drug: bimatoprost vehicle solution
- minoxidil 2% solution (Active Comparator): Approximately one mL dose applied evenly onto pre-specified area on scalp, twice daily for 6 months.
  Interventions: Drug: minoxidil 2% solution

INTERVENTIONS:
Drug: bimatoprost Formulation A — Approximately one mL dose applied evenly onto pre-specified area on scalp, once daily for 6 months.
  Arms: bimatoprost Formulation A
Drug: bimatoprost Formulation B — Approximately one mL dose applied evenly onto pre-specified area on scalp, once daily for 6 months.
  Arms: bimatoprost Formulation B
Drug: bimatoprost Formulation C — Approximately one mL dose applied evenly onto pre-specified area on scalp, once daily for 6 months.
  Arms: bimatoprost Formulation C
Drug: bimatoprost vehicle solution — Approximately one mL dose applied evenly onto pre-specified area on scalp, once daily for 6 months.
  Arms: bimatoprost vehicle solution
Drug: minoxidil 2% solution — Approximately one mL dose applied evenly onto pre-specified area on scalp, twice daily for 6 months.
  Other Names: Rogaine®; Regaine®
  Arms: minoxidil 2% solution

SUMMARY:
This study will evaluate the safety and efficacy of 3 doses of bimatoprost solution compared with vehicle and over-the-counter (OTC) minoxidil 2% solution in women with female pattern hair loss. All treatments will be provided in a double-blinded fashion except for minoxidil 2% solution which will be provided open-label.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate female pattern hair loss with ongoing hair loss for at least 1 year
* Willingness to have micro-dot-tattoo applied to scalp
* Willingness to maintain same hair style, length and hair color during study

Exclusion Criteria:

* Drug or alcohol abuse within 12 months
* HIV positive
* Received hair transplants or had scalp reductions
* Use of hair weaves, hair extensions or wigs within 3 months
* Oral or topical minoxidil treatment within 6 months
* Application of topical steroids or nonsteroidal anti-inflammatory drugs (NSAIDs) to scalp within 4 weeks

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 306 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Portland, Oregon, United States
- Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Bimatoprost Formulation A: Approximately one milliliter (mL) of bimatoprost Formulation A applied evenly onto pre-specified area on scalp, once daily for 6 months.
- Bimatoprost Formulation B: Approximately one mL of bimatoprost Formulation B applied evenly onto pre-specified area on scalp, once daily for 6 months.
- Bimatoprost Formulation C: Approximately one mL of bimatoprost Formulation C applied evenly onto pre-specified area on scalp, once daily for 6 months.
- Vehicle to Bimatoprost: Approximately one mL of vehicle to bimatoprost applied evenly onto pre-specified area on scalp, once daily for 6 months.
- Minoxidil 2% Solution: Approximately one mL of minoxidil 2% solution applied evenly onto pre-specified area on scalp, twice daily for 6 months.
Period: Overall Study
Arm/Group | Bimatoprost Formulation A | Bimatoprost Formulation B | Bimatoprost Formulation C | Vehicle to Bimatoprost | Minoxidil 2% Solution
Started | 61 | 61 | 61 | 61 | 62
Completed | 55 | 56 | 44 | 52 | 50
Not Completed | 6 | 5 | 17 | 9 | 12
Not completed — Adverse Event | 3 | 3 | 3 | 1 | 2
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 5 | 1 | 5
Not completed — Personal Reasons | 2 | 1 | 6 | 5 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0
Not completed — Did Not Receive Treatment | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bimatoprost Formulation A: Approximately one mL of bimatoprost Formulation A applied evenly onto pre-specified area on scalp, once daily for 6 months.
- Total: Total of all reporting groups
Arm/Group | Bimatoprost Formulation A | Bimatoprost Formulation B | Bimatoprost Formulation C | Vehicle to Bimatoprost | Minoxidil 2% Solution | Total
Number analyzed (Participants) | 61 | 61 | 61 | 61 | 62 | 306
Age, Customized [Number; unit: Participants]
  18 to 34 years | 12 | 13 | 12 | 13 | 12 | 62
  35 to 59 years | 49 | 48 | 49 | 48 | 50 | 244
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 61 | 61 | 61 | 62 | 306
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Target Area Hair Count (TAHC)
Description: TAHC was measured using digital imaging analysis and was reported in terminal hairs/centimeters squared (cm^2). A positive change from Baseline indicated improvement (increase in the number of terminal hairs). A negative change from Baseline indicated worsening (decrease in the number of terminal hairs).
Time Frame: Baseline, Month 6
Population: Participants from the Modified Intent-to-Treat Population (all randomized participants who received treatment and had both Baseline and post-Baseline measurements) who had data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: terminal hairs/cm^2
Arm/Group | Bimatoprost Formulation A | Bimatoprost Formulation B | Bimatoprost Formulation C | Vehicle to Bimatoprost | Minoxidil 2% Solution
Number analyzed (Participants) | 61 | 60 | 60 | 61 | 61
terminal hairs/cm^2
  Baseline | 153.1 (54.78) | 161.1 (63.85) | 145.2 (63.42) | 163.0 (57.28) | 156.3 (55.46)
  Change from Baseline at Month 6 | -0.4 (17.10) | -3.5 (18.21) | 4.3 (16.82) | 1.1 (20.44) | 13.6 (18.72)

2. Primary Outcome: Percentage of Participants in Each Response Category of the Subject Self Assessment in Alopecia (SSA) Score
Description: The SSA score measured scalp hair growth. Using a 7-point scale, participants answered the Question: "Since the start of the study, the amount of my hair has?": Greatly Increased, Moderately Increased, Slightly Increased, Remained the Same, Slightly Decreased, Moderately Decreased or Greatly Decreased. The percentage of participants in each response category is presented.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost Formulation A | Bimatoprost Formulation B | Bimatoprost Formulation C | Vehicle to Bimatoprost | Minoxidil 2% Solution
Number analyzed (Participants) | 58 | 60 | 54 | 61 | 56
Percentage of participants
  Greatly Increased | 3.4 | 3.3 | 9.3 | 3.3 | 7.1
  Moderately Increased | 17.2 | 20.0 | 16.7 | 18.0 | 28.6
  Slightly Increased | 34.5 | 21.7 | 16.7 | 24.6 | 35.7
  Remained the Same | 20.7 | 33.3 | 38.9 | 29.5 | 19.6
  Slightly Decreased | 19.0 | 11.7 | 13.0 | 13.1 | 5.4
  Moderately Decreased | 1.7 | 8.3 | 5.6 | 8.2 | 1.8
  Greatly Decreased | 3.4 | 1.7 | 0.0 | 3.3 | 1.8

3. Secondary Outcome: Percentage of Participants in Each Response Category of the Investigator Global Assessment (IGA) Score
Description: The investigator compared the participant's scalp hair growth at Month 6 to a photograph of the scalp taken at Baseline and using the 7-point IGA score, the investigator answered the question: "Since the start of the study, the amount of the subject's hair has?": Greatly Increased, Moderately Increased, Slightly Increased, Remained the Same, Slightly Decreased, Moderately Decreased or Greatly Decreased. The percentage of participants in each response category is presented.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost Formulation A | Bimatoprost Formulation B | Bimatoprost Formulation C | Vehicle to Bimatoprost | Minoxidil 2% Solution
Number analyzed (Participants) | 58 | 60 | 54 | 61 | 56
Percentage of participants
  Greatly Increased | 5.2 | 3.3 | 7.4 | 1.6 | 1.8
  Moderately Increased | 12.1 | 10.0 | 11.1 | 14.8 | 16.1
  Slightly Increased | 24.1 | 35.0 | 25.9 | 23.0 | 37.5
  Remained the Same | 39.7 | 40.0 | 51.9 | 54.1 | 41.1
  Slightly Decreased | 15.5 | 10.0 | 3.7 | 6.6 | 3.6
  Moderately Decreased | 3.4 | 1.7 | 0.0 | 0.0 | 0.0
  Greatly Decreased | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Percentage of Participants in Each Response Category of the Global Panel Review (GPR) Score
Description: At the completion of the study, 3 independent dermatologists using the 7-point GPR score compared photographs of the participant's scalp hair growth at Month 6 to Baseline and answered the question: "Compared with the baseline image, the amount of the subject's hair has?": Greatly Increased, Moderately Increased, Slightly Increased, Remained the Same, Slightly Decreased, Moderately Decreased or Greatly Decreased. The percentage of participants in each response category is presented.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Bimatoprost Formulation A | Bimatoprost Formulation B | Bimatoprost Formulation C | Vehicle to Bimatoprost | Minoxidil 2% Solution
Number analyzed (Participants) | 55 | 59 | 48 | 61 | 53
Percentage of participants
  Greatly Increased | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Moderately Increased | 1.8 | 0.0 | 2.1 | 1.6 | 0.0
  Slightly Increased | 0.0 | 6.8 | 6.3 | 6.6 | 17.0
  Remained the Same | 87.3 | 81.4 | 81.3 | 88.5 | 79.2
  Slightly Decreased | 10.9 | 11.9 | 10.4 | 3.3 | 1.9
  Moderately Decreased | 0.0 | 0.0 | 0.0 | 0.0 | 1.9
  Greatly Decreased | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

5. Secondary Outcome: Change From Baseline in Target Area Hair Width (TAHW)
Description: Digital imaging analysis was used to measure TAHW in millimeters/centimeters squared (mm/cm^2). The diameters of all terminal hairs (individual hairs ≥ 30 microns) in the target area were summed and reported together. A positive change from Baseline indicated improvement (increase in the diameter of terminal hairs). A negative change from Baseline indicated worsening (decrease in the diameter of terminal hairs).
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/cm^2
Arm/Group | Bimatoprost Formulation A | Bimatoprost Formulation B | Bimatoprost Formulation C | Vehicle to Bimatoprost | Minoxidil 2% Solution
Number analyzed (Participants) | 61 | 60 | 60 | 61 | 61
mm/cm^2
  Baseline | 8.92 (3.444) | 9.64 (3.308) | 8.86 (3.977) | 10.13 (4.165) | 9.76 (3.698)
  Change from Baseline from Month 6 | 0.13 (1.198) | -0.19 (1.067) | 0.30 (1.263) | 0.07 (1.183) | 0.87 (1.315)

6. Secondary Outcome: Change From Baseline in Target Area Hair Darkness (TAHD)
Description: Digital imaging analysis was used to measure TAHD. The darkness of all terminal hairs (individual hairs ≥ 30 microns) in the target area were summed and divided by total number of terminal hairs in the same target area and was reported as intensity units. A positive change from Baseline indicated improvement (increase in the darkness of terminal hairs).
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Intensity units
Arm/Group | Bimatoprost Formulation A | Bimatoprost Formulation B | Bimatoprost Formulation C | Vehicle to Bimatoprost | Minoxidil 2% Solution
Number analyzed (Participants) | 61 | 60 | 60 | 61 | 61
Intensity units
  Baseline | 95.63 (23.837) | 100.12 (25.077) | 92.76 (19.433) | 96.90 (22.678) | 93.07 (20.667)
  Change from Baseline at Month 6 | 2.94 (13.084) | 4.22 (13.159) | 2.11 (14.674) | 2.07 (11.486) | 2.12 (11.561)

ADVERSE EVENTS:
Description: The Safety Population (all participants who received at least 1 dose of study treatment) was used to calculate the number of participants at risk for treatment-emergent Serious Adverse Events and treatment-emergent Adverse Events.
Arm/Group | Bimatoprost Formulation A | Bimatoprost Formulation B | Bimatoprost Formulation C | Vehicle to Bimatoprost | Minoxidil 2% Solution
Serious Adverse Events (participants affected / at risk) | 4/61 | 4/60 | 3/60 | 1/61 | 1/61
Other Adverse Events (participants affected / at risk) | 17/61 | 17/60 | 15/60 | 20/61 | 24/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Formulation A (N=61) | Bimatoprost Formulation B (N=60) | Bimatoprost Formulation C (N=60) | Vehicle to Bimatoprost (N=61) | Minoxidil 2% Solution (N=61)
Death (General disorders) | 0 | 0 | 1 | 0 | 0 — Event not treatment-related
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 — Event not treatment-related
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 — Event not treatment-related
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 — Event not treatment-related
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 — Events not treatment-related
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 — Event not treatment-related
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 — Event not treatment-related
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 — Events not treatment-related
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 — Event not treatment-related
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 — Event not treatment-related
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 — Event not treatment-related
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 — Event not treatment-related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost Formulation A (N=61) | Bimatoprost Formulation B (N=60) | Bimatoprost Formulation C (N=60) | Vehicle to Bimatoprost (N=61) | Minoxidil 2% Solution (N=61)
Application site pruritis (General disorders) | 0 | 3 | 2 | 0 | 5
Application site dryness (General disorders) | 1 | 1 | 0 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 6 | 7
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 4 | 5 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 1 | 3
Hypertension (Vascular disorders) | 0 | 0 | 3 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 3 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.